CLINICAL TRIAL: NCT01102582
Title: A Six-month Observational Study to Investigate Prevalence of Neuropsychiatric Symptom in Korean Patients With Parkinson's Disease Dementia
Brief Title: An Observational Study for the Prevalence of Neuropsychiatric Symptom in Parkinson's Disease Dementia
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Collaborators: Yonsei University (Other)
Responsible Party: Principal Investigator, Joong-Seok Kim, Professor, The Catholic University of Korea
Other Study IDs: Norva100408
Record Dates: First submitted 2010-04-08; First posted 2010-04-13 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Parkinson's Disease Dementia
Keywords: Parkinson's disease dementia, neuropsychiatric symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
* Dementia correlates to decreased cognitive function, and Behavioral and Psychological Symptoms of Dementia (Neuropsychiatric symptom, BPSD) as well.
* Neuropsychiatric symptom attributes important role for mortality, mortality, and cause to enter nursing home.
* Study on neuropsychiatric symptom in patients with Parkinson's disease has not been thorough yet, and there even has not been any study done on this in Korea yet.
* The investigators will study prevalence of neuropsychiatric symptom in PDD patients and burden of caregiver.

DETAILED DESCRIPTION:
* It is well recognized that the importance of non-motor symptoms of Parkinson's disease during its progression and many patients are suffering from this. The deterioration of cognitive function is especially known as a crucial prognostic factor. According to recently released cohort study, majority of patients go through dementia in advanced Parkinson's disease.
* Dementia correlates to decreased cognitive function, and Behavioral and Psychological Symptoms of Dementia (Neuropsychiatric symptom, BPSD) as well. Neuropsychiatric symptom composed of abnormal behavior and psychological symptoms: abnormal behaviors include combativeness, wandering, agitation, akathisia, inappropriate sexual behavior, following caregiver, shouting, cursing, insomnia and binge eating while psychological symptoms include anxiety, depression, hallucination, and illusion. Neuropsychiatric symptom is evaluated depending on information given by caregivers, and symptoms are likely to be temporary or changing constantly. Two thirds of patients is found to have neuropsychiatric symptom when they are diagnosed as dementia, 65 % in nursing home and 70~90% in advanced dementia states. Neuropsychiatric symptom attributes important role for mortality, mortality, and cause to enter nursing home.
* Besides, neuropsychiatric symptom also plays important part as care-giver burden. It gives heavier burden on caregiver rather than on patients, and increases depression and anxiety of caregivers. Specific correlation with patient's neuropsychiatric symptom to burden of caregiver is known as agitation, depression, aggression, repetitive behavior, anxiety, and disinhibition. There are, however, various results related to race, region, subjects, and investigator.
* Study on neuropsychiatric symptom in patients with Parkinson's disease dementia has not been thorough yet, and there even has not been any study done on this in Korea yet.
* The investigators will study prevalence of neuropsychiatric symptom in PDD patients and burden of caregiver.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed of Parkinson's disease dementia.
* Written informed consent will be obtained from the patient (if possible) or from the patient's legal guardian or other representative prior to beginning the any baseline assessments or activities. Even if unable to provide written informed consent, the patient must assent verbally to participating in the study.
* The regimen for levodopa that was administered regularly to patients for 1 month before the enrollment can be adjusted optimally for the patients during the investigation.
* Patients with other dopamine enhancer, MAO-B inhibitor or Amantadine administered should be kept stable state during this study.
* Patients who have been on other medication for 1 month before they are enrolled can be included if the investigator decides that those medication won't affect the result of the study.
* Other medication for the treatment of other disease can be administered under discussion with the physician in charge or those medications.

Exclusion Criteria:

* Patients who are under other study.
* Patients with other systemic disease who are to be limited for drug administration.
* Patients who are pregnant.
* Participants are not allowed to take any other medication that can affect cognitive function e.g, anti-cholinergic medications, benztropine, trihexphenidyl, and biperidene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The tertiary clinic in university hospital
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric inventory | Baseline
  It collects information on symptoms during the past month in 10 domains-delusions, hallucinations, agitation, depression, anxiety, elation, apathy, disinhibition, irritability, and aberrant motor behaviors-using a structured interview with a knowledgeable informant.

SECONDARY OUTCOMES:
Follow-up neuropsychiatric inventory | Six months after choline esterase inhibitor treatment
  The change of prevalence of neuropsychiatric symptoms after choline esterase inhibitor treatment.
Care-giver burden_baseline | Baseline
  The burden of caregiver determined by Burden Interview(BI) and Caregiver Burden inventory(CBI)
Care-giver burden change | Six months after choline esterase inhibitor treatment
  The burden change of caregiver using the same scale (BI and CBI).
Motor function_baseline | Baseline
  Hoehn and Yahr stage and Unified Parkinson's disease rating scale, part 3
Motor function_change | Six months after choline esterase inhibitor treatment
  Hoehn and Yahr stage and Unified Parkinson's Disease Rating Scale
General cognitive function_baseline | Baseline
  The Korean version of mini mental status examination, clinical dementia rating, Barthel and Instrumental ADL
General cognitive function_change | Six months after choline esterase inhibitor treatment
  The Korean version of mini mental status examination, clinical dementia rating, Barthel and Instrumental ADL

CONTACTS AND LOCATIONS:
Overall Officials: Joong-Seok Kim, MD, Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea, Yonsei University, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Aarsland D, Cummings JL, Larsen JP. Neuropsychiatric differences between Parkinson's disease with dementia and Alzheimer's disease. Int J Geriatr Psychiatry. 2001 Feb;16(2):184-91. doi: 10.1002/1099-1166(200102)16:23.0.co;2-k. PMID 11241724
- [Background] Aarsland D, Bronnick K, Ehrt U, De Deyn PP, Tekin S, Emre M, Cummings JL. Neuropsychiatric symptoms in patients with Parkinson's disease and dementia: frequency, profile and associated care giver stress. J Neurol Neurosurg Psychiatry. 2007 Jan;78(1):36-42. doi: 10.1136/jnnp.2005.083113. Epub 2006 Jul 4. PMID 16820421